CLINICAL TRIAL: NCT02638025
Title: Anterior Segment Spectral-domain Optical Coherence Tomography in Patients With Closed Globe Injury
Status: Completed | Type: Observational
Sponsor: Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HMCH20151216
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Eye Injuries
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: OCT — Anterior Segment Spectral-domain Optical Coherence Tomography

SUMMARY:
This study use anterior segment spectral-domain optical coherence tomography (SD-OCT) to exam patients with closed globe injury, and compared with slit lamp examination. The results showed that OCT can identify features of closed globe injury that were otherwise not visible on slit lamp biomicroscopy.

DETAILED DESCRIPTION:
The anterior segment architecture changes of closed globe injury patients include corneal damage, hyphema, angle recession and lens dislocation, which can be showed with OCT. OCT was superior to slit lamp biomicroscopy examination in detecting anterior segment architecture changes, especially in the presence of media opacities.

ELIGIBILITY:
Inclusion Criteria:

* patients with closed globe injury were recruited; had hyphema at least 1/3 of anterior chamber volume

Exclusion Criteria:

* can not cooperate with examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with closed globe injury were recruited, and all eyes of recruited patients had hyphema occupying at least 1/3rd of anterior chamber volume
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
anterior segment spectral-domain optical coherence tomography (SD-OCT) findings in patients with closed globe injury | within 24 hours after patients were admitted